CLINICAL TRIAL: NCT01367938
Title: OMNI Apex Knee Ultracongruent vs. Triathlon® Posterior Stabilized & Cruciate Substituting Outcomes Study
Brief Title: Clinical Outcomes With Omni Apex Ultracongruent Knee System
Status: Completed | Type: Observational
Sponsor: Spokane Joint Replacement Center (Other)
Responsible Party: Principal Investigator, David F. Scott, MD, PI, Spokane Joint Replacement Center
Other Study IDs: SJRC-OK
Record Dates: First submitted 2011-05-22; First posted 2011-06-07 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Total Knee Replacement; Total Knee Arthroplasty; TKA; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- OMNI Apex Ultracongruent Knee Device
  Interventions: Device: OMNI Apex Ultracongruent Knee Device

INTERVENTIONS:
Device: OMNI Apex Ultracongruent Knee Device

SUMMARY:
A prospective, matched case comparison of total knee arthroplasty with the OMNI Apex Ultracongruent vs. Triathlon® CS tibial insert vs. the Triathlon® PS tibial insert.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to sign the informed consent.
* Patients able to comply with follow-up requirements including postoperative weight bearing restrictions and self-evaluations.
* Male and non-pregnant female patients ages 21-80 years of age at time of surgery.
* Patients requiring a primary total knee replacement.
* Patients with a diagnosis of osteoarthritis (OA), traumatic arthritis (TA), or avascular necrosis (AVN).
* Patients with intact collateral ligaments.

Exclusion Criteria:

* Patients with inflammatory arthritis.
* Patients that are morbidly obese, body mass index (BMI) > 40.
* Patients with a history of total or unicompartmental reconstruction of the affected joint.
* Patients that have had a high tibial osteotomy or femoral osteotomy.
* Patients with neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
* Patients with a systemic or metabolic disorder leading to progressive bone deterioration.
* Patients that are immunologically compromised, or receiving chronic steroids (>30 days).
* Patients bone stock is compromised by disease or infection, which cannot provide adequate support and/or fixation to the prosthesis.
* Patients with knee fusion to the affected joint.
* Patients with an active or suspected latent infection in or about the knee joint.
* Patients that computer-assisted surgical navigation (CAOS) techniques will be used.
* Patients that minimally invasive surgical technique will be used.
* Patients that are prisoners.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing total knee replacement
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2009-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes | Pre-operative, 6 weeks, 6 months, 1, 2, 3, 4, and 5 years post-operative
  Clinical outcomes to include overall success, revision rate, adverse events, clinical score (Knee Society Score), range of motion, radiographic findings.

CONTACTS AND LOCATIONS:
Overall Officials: David F Scott, MD, Principal Investigator — Spokane Joint Replacement Center
Locations (1):
- Spokane Joint Replacement Center, Spokane, Washington, United States